CLINICAL TRIAL: NCT02175381
Title: A Phase I/II Trial of the Carboplatin/Gemcitabine Combination as First Line Treatment for Elderly Patients With Stage IV NSCLC.
Brief Title: Carboplatin Plus Gemcitabine for Elderly Patients With Stage IV NSCLC
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/10.04
Record Dates: First submitted 2014-06-21; First posted 2014-06-26 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: NSCLC
Keywords: Metastatic NSCLC; Elderly; 1st Line; Platinum-based treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carbo/GEM (Experimental)
  Interventions: Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Carboplatin — Carboplatin: 2.5 AUC i.v on day 1. Cycle repeated ever 2 weeks
Drug: Gemcitabine — Gemcitabine: 1100 mg/m2, iv on day 1. Cycle repeated every 2 weeks

SUMMARY:
The investigators propose to study the safety and efficacy of the combination of Carboplatin plus Gemcitabine in a Phase I/II trial of elderly subjects with non-small cell lung cancer.

DETAILED DESCRIPTION:
About 50% of newly diagnosed cases of NSCLC concern patients older than 65 years, while 30-40% of cases are diagnosed in patients older than 70 years. Furthermore, recent data suggest that during the last decade, the incidence and mortality of NSCLC has decreased in younger patients, while it has increased among older patients. Based on these observations, it becomes clear that NSCLC represents a significant health problem in elderly patients. However, elderly patients are frequently underrepresented in clinical trials evaluating new treatments in NSCLC. Indeed, more than 75% of patients older than 65 years with metastatic NSCLC never receive any kind of chemotherapy in the daily clinical practice.

In elderly patients there is lack of prospective data regarding the role of platinum-based doublets. It is not clear whether elderly patients gain any survival benefit or not from platinum-based doublets and whether these chemotherapeutic regimens result in a significant increase in toxicity.

There is a clear need to prospectively evaluate the tolerability and efficacy of platinum-based doublets as first-line chemotherapy for older NSCLC patients.

On this basis it would be very interesting to initiate a phase I/II study with gemcitabine/carboplatin combination as first line treatment in older NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥70 years old
* Cytologically or histologically documented NSCLC
* Measurable disease according to Response Evaluation Criteria in Solid Tumors (at least one measurable lesion)
* World Health Organisation (WHO) performance status 0-2
* Non-frail patients according to Comprehensive Geriatric Assessment
* Previously treated NSCLC (or patients for whom the combination is considered adequate treatment) (for phase I part)
* No prior chemotherapy (for phase II part)
* Life expectancy of at least 12 weeks
* Serum bilirubin less than 1.5 times the upper normal limit
* Aspartate Aminotransferase and Alanine Aminotransferase less than 2.5 times the upper normal limit in the absence of demonstrable liver metastases, or less than 5 times the upper normal limit in the presence of liver metastases
* Serum creatinine less than 1.5 times the upper normal limit and Creatinine Clearance >60 ml/min
* Neutrophil count more than 1.5x 109 /L
* Platelet count more than 100x 109 /L
* Before patient enrollment, written informed consent must be given according to Good Clinical Practice guidelines and national/local regulations.

Exclusion Criteria:

* Hemoptysis
* Central nervous system metastases
* Clinically significant cardiovascular disease
* Medically uncontrolled hypertension
* Other co-existing malignancies or malignancies diagnosed within the last 5 years (with the exception of basal cell carcinoma or cervical cancer in situ)
* Any evidence of severe uncontrolled concomitant disease (in the opinion of the investigator)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Disease evaluation at Week 8

SECONDARY OUTCOMES:
Disease control rate | Disease evaluation at Week 8
  Disease control rate is defined as the proportion of patients with complete response or partial response or stable disease for at least 16 weeks
Progression Free Survival | 1 year
Overall Survival | 1 year
Safety Profile | Every two weeks up to 12 weeks
  Patients will be evaluated for Adverse Events (related or unrelated to the treatment) on Day 1 of each cycle (cycle repeated every 2 weeks) up to 12 weeks from the date of first dose administration

CONTACTS AND LOCATIONS:
Overall Officials: Lambros Vamvakas, MD, Principal Investigator — University Hospital of Herklion; Athanasios Karambeazis, MD, Principal Investigator — Medical Oncology Unit NIMTS (Veterans Hospital)
Locations (5):
- Greece (5):
  - University Hospital of Crete, Dep of Medical Oncology Heraklion, Greece, Heraklion, Crete
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - 401 Military Hospital of Athens, Athens
  - Air Forces Military Hospital of Athens Athens, Greece, Athens
  - Medical Oncology Unit NIMTS (Veterans Hospital), Athens